CLINICAL TRIAL: NCT00937014
Title: Assessment of Growth of Infants Fed a Starter Formula With a Whey-Isolate Enriched in Lactoferrin
Brief Title: Assessment of Growth of Infants Fed a New Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 07.35.INF
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Infant Nutrition
Keywords: infant formula; growth; weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard infant formula (Active Comparator)
  Interventions: Other: standard infant formula
- Test formula (Experimental)
  Interventions: Other: Test formula

INTERVENTIONS:
Other: standard infant formula — Standard infant formula given during the first 9 months of life, as per standard requirement
  Arms: Standard infant formula
Other: Test formula — Test formula enriched in lactoferrin given during the first 9 months of life, as per standard requirement.
  Arms: Test formula

SUMMARY:
The purpose of this clinical trial is to assess growth (rate of weight gain in grams per day) of infants fed an infant formula with a whey isolate enriched with lactoferrin, during the first four months of life as compared to infants fed a standard infant formula.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infant
* Full-term (>37 weeks gestation)
* Birth weight between > 2500 and < 4500 g
* Infant's mother has elected not to breastfeed and baby has been exclusively formula fed a minimum 3 days prior to enrollment
* Tolerating a cows milk based formula for at least 3 days
* Study explained and written information provided with Parent/Caregiver demonstrating understanding of the given information
* Informed consent signed (Parent/Legal representative)
* Parent/Caregiver has a working freezer
* Lives within 45 minutes of a study site

Exclusion Criteria:

* Congenital illness or malformation that may affect infant feeding and/or normal growth
* Suspected or known allergy to cow's milk protein
* Significant pre-natal and/or post-natal disease
* Any readmission to hospital (except for hyperbilirubinemia) prior to enrollment
* Infant has received oral or intravenous antibiotic therapy in the 10 days prior to enrollment
* Infant receiving prescription medication (with exception of treatment for thrush) or frequent use of over the counter medications except vitamin and mineral supplements
* Infant currently participating in another clinical study
* Infant's family who in the Investigator's assessment cannot be expected to comply with the protocol

Ages: 11 Days to 17 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Mean weight gain | 4 months

SECONDARY OUTCOMES:
anthropometry, tolerance, morbidity, blood tests | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan Feigelman, MD, Principal Investigator — University of Maryland School of Medicine, Department of Pediatrics
Locations (3):
- United States (3):
  - Pedia Research, LLC, Newburgh, Indiana
  - Pedia Research, LLC, Owensboro, Kentucky
  - University of Maryland School of Medicine, Baltimore, Maryland